CLINICAL TRIAL: NCT03919656
Title: SGLT-2 Inhibition and Cardiovascular Disease. Metabolomics Study of Potential Factors Involved in Cardio- and Nephroprotection
Brief Title: SGLT-2 Inhibition, Metabolomics and Cardiovascular/Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FIM-DAPA-2018-01
Record Dates: First submitted 2019-04-11; First posted 2019-04-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metabolomics; Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Who Masked: Participant, Investigator
Masking Description: Dapagliflozin 10 mg, Green, plain, diamond shaped, film coated tablet (orally); Matching placebo for dapagliflozin Green, plain, diamond shaped, film coated tablet (orally). Does not contain active ingredient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg daily (orally)
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator): Matching placebo for dapagliflozin daily (orally). Does not contain active ingredient
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Dapagliflozin 10 mg daily in a green, plain, diamond shaped, film coated tablet (orally)
  Other Names: Farxiga 10 mg
  Arms: Dapagliflozin
Drug: Placebo Oral Tablet — Green, plain, diamond shaped, film coated tablet (orally). Does not contain active ingredient
  Arms: Placebo

SUMMARY:
This study evaluates the metabolomics changes associated with dapagliflozin treatment in patients with type 2 diabetes mellitus (T2DM). The participants in the study will be randomized to receive 10 mg dapagliflozin or placebo once daily for 12 weeks.

DETAILED DESCRIPTION:
In this study, we hypothesize that metabolomics changes that occur in patients with T2DM after initiating SGLT2i (sodium-glucose cotransporter 2 inhibitors) treatment may be responsible for the beneficial cardiovascular and kidney effects observed in clinical trials with SGLT2i. Also, we propose that the study of the specific metabolome associated with the treatment with SGLT2i could help identify the possible metabolites and molecules that reduce CVD (cardiovascular disease) and renal disease in patients with T2DM.

The participants in the study will be randomized to receive 10 mg dapagliflozin or placebo once daily of for 12 weeks. Besides, all participants will be advised to engage in 150 min or more of moderate-to vigorous intensity physical activity per week, spread over at least 3 days/week, with no more than 2 consecutive days without activity and to engage in 2-3 sessions/week of resistance exercise on nonconsecutive days. Moreover, these patients will be advised to follow a lifestyle program that achieve a 500-750 kcal/day energy deficit or provide≈1,200-1,500 kcal/day for women and 1,500-1,800 kcal/day for men, adjusted for the individual's baseline body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75.
* BMI 27-39.9 kg/m2.
* T2DM on treatment with metformin and inadequate metabolic control (defined as HbA1c≥6.5 -7%).

Exclusion Criteria:

* Pregnancy (all women of child-bearing age, unless on treatment with contraceptive methods, will undergo a pregnancy test)
* Breastfeeding
* Intolerance/allergy to dapagliflozin.
* Treatment with antidiabetic drug other than metformin.
* Impaired kidney function: Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 (calculated using the CKD-EPI formula).
* Patients with established cardiovascular disease.
* Previous or current history of cancer of any kind.
* Uncontrolled hypertension (systolic blood pressure≥160 mmHg or diastolic blood pressure≥110 mmHg, despite adequate antihypertensive treatment).
* History of liver tumour or acute or chronic liver disease with impaired liver function: total bilirubin levels> 2.0 mg / dl or GOT/GPT levels three times higher than normal upper limit.
* Known HIV infection or active HBV or HCV infection.
* Other serious underlying diseases, which could affect the patient's ability to participate in the study.
* Reduced life expectancy (<12 months) due to advanced or terminal concomitant diseases.

In addition, female patients of child-bearing age will be advised to use contraceptive methods during the study period, given the contraindication of dapagliflozin and metformin during pregnancy as per normal clinical practice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Metabolomics changes in blood | From baseline to week 12
  Targeted and quantitative analysis by ultra-high-resolution liquid chromatography coupled to triple quadrupole mass spectrometry (UHPL-QqQ/MS). Analysis of specific families of metabolites selected from hypotheses generated by previous exploratory studies: changes in acylcarnitines and other intermediates of mitochondrial β-oxidation and the urea cycle, branched-chain amino acids and biogenic amines
Metabolomics changes in urine | From baseline to week 12
  Targeted and quantitative analysis by ultra-high-resolution liquid chromatography coupled to triple quadrupole mass spectrometry (UHPL-QqQ/MS). Analysis of specific families of metabolites selected from hypotheses generated by previous exploratory studies: changes in acylcarnitines and other intermediates of mitochondrial β-oxidation and the urea cycle, branched-chain amino acids and biogenic amines

SECONDARY OUTCOMES:
BMI (body mass index) changes | From baseline to to week 12
  Measured by body composition analysis
Changes in insulin resistance | From baseline to to week 12
  Measured as HOMA-IR (homeostatic model assessment of insulin resistance)
Changes in metabolic control | From baseline to to week 12
  Measured as HbA1c (glycated hemoglobin)
Changes in Quality of Life: 36-Item Short Form Health Survey (SF-36) questionnaire | From baseline to to week 12
  The SF-36 has eight scaled scores: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The scores are weighted sums of the questions in each section. Scores range from 0 - 100, lower scores indicate more disability, and higher scores indicate less disability
Changes in albuminuria | From baseline to to week 12
  Modifications in albuminuria, measured as albumin excretion rate (AER)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos Fernandez-Garcia, MD, PhD, Principal Investigator — Virgen de la Victoria Hospital
Locations (1):
- Virgen de la Victoria University Hospital. Endocrinology Department, Málaga, Spain, Spain

IPD SHARING:
Plan to Share IPD: No